CLINICAL TRIAL: NCT04477317
Title: Anesthetic Efficacy of %4Alexadricaine Versus %2 Mepicaine-L for Infiltration Anesthesia in Extraction of Maxillary First Primary Molars in Children
Brief Title: Anesthetic Efficacy of %4Alexadricaine Versus %2 Mepicaine-L in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Mostafa Mahmoud, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: local anesthesia in chilldren
Record Dates: First submitted 2020-07-13; First posted 2020-07-20 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Local Anesthesia
MeSH Terms: interventions — Carticaine; Epinephrine; Mepivacaine; Nordefrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): 4% Articaine Hydrochloride with 1:100,000 Adrenaline (Alexadricaine, Alexandria Co., Egypt).
  Interventions: Drug: 4% Articaine Hydrochloride with 1:100,000 Adrenaline
- Control (Active Comparator): 2% Mepivacaine Hydrochloride with 1:20,000 Levonordefrin (Mepicaine-L, Alexandria Co., Egypt)
  Interventions: Drug: 2% Mepivacaine Hydrochloride with 1:20,000 Levonordefrin

INTERVENTIONS:
Drug: 4% Articaine Hydrochloride with 1:100,000 Adrenaline — new Egyptian articane anesthetic solution.
  Other Names: %4 Alexadricaine
  Arms: Experimental
Drug: 2% Mepivacaine Hydrochloride with 1:20,000 Levonordefrin — Mepecaine-L is the brand name of the Egyptian 2% Mepivacaine. It is the most commonly used anesthetic solution in Egypt due to its availability and its lower cost.
  Other Names: 2% Mepicaine-L
  Arms: Control

SUMMARY:
The aim of the present study is to evaluate and compare the anesthetic efficacy of Alexadricaine versus Mepecaine-L infiltration anesthesia in children during extraction of badly decayed or unrestorable maxillary first primary molars.

DETAILED DESCRIPTION:
To our knowledge, no clinical trials in literature have been done to compare anesthetic efficacy of 4% Articaine versus 2% Mepivacaine in pain management during extraction of badly decayed upper first primary molars. Thus, the purpose of the present study was to fill this knowledge gap.

This trial will be held on a new brand of 4% articaine made in Egypt called Alexadricaine anesthetic solution where no clinical trials have been conducted on it yet in literature.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit (ASA I, II).
* Mentally capable of communication.
* Children aged 5-7 years, children older than 8 years old will not be included due to physiologic root resorption associated with shedding which may simplify the extraction procedure(25).
* First maxillary primary molar needs extraction due to root caries "beyond possible repair".
* First dental visit.
* Child must give assent prior to participation, as well as approved parental informed written consent.

Exclusion Criteria:

* Children with acute or sub-acute dento-alveolar abscess Children with history of prolonged bleeding, platelet disorders, Hyperthyroidism or hypersensitivity.
* Patients who had taken analgesics or antibiotics in the 12-hrs preceding the injection.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Intra-operative pain during extraction | through study completion, an average of 1 year
  measured by Visual Analogue Scale (VAS) and Sound Eye Motor (SEM) scale

SECONDARY OUTCOMES:
onset of anesthesia | through study completion, an average of 1 year
  measured in minutes using stopwatch
duration of anesthesia | through study completion, an average of 1 year
  measured in minutes using stopwatch

CONTACTS AND LOCATIONS:
Overall Officials: Sara A mahmoud, Assoc. Prof., Study Director — Cairo University
Locations (1):
- Faculty of dentistry cairo university, Cairo, Egypt